CLINICAL TRIAL: NCT00634322
Title: Randomized, Blinded, Placebo-Controlled Trial of High Dose Methotrexate With Leucovorin Rescue (HDMTX-LV) With or Without Glucarpidase in Osteosarcoma
Brief Title: High Dose Methotrexate With Leucovorin Rescue With or Without Glucarpidase in Osteosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: BTG International Inc. (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR001-CLN-pro012; MDACC #2006-0246
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; high dose methotrexate; leucovorin
MeSH Terms: conditions — Osteosarcoma | interventions — glucarpidase; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): HDMTX-LV with glucarpidase
  Interventions: Drug: glucarpidase
- B (Active Comparator): HDMTX-LV with placebo
  Interventions: Drug: leucovorin
- C (Experimental): compassionate use group to treat or prevent life threatening toxicity in the event of delayed elimination of MTX and/or renal impairment
  Interventions: Drug: glucarpidase

INTERVENTIONS:
Drug: glucarpidase — IV dose based on weight, two doses given for 5 minutes, 24 hours apart
  Other Names: Voraxaze, caboxypeptidase G2, CPG2
  Arms: A; C
Drug: leucovorin — IV or po given every 6 hours
  Other Names: LV
  Arms: B

SUMMARY:
The purpose of this study is to demonstrate whether use of glucarpidase facilitates administration of the next cycle of chemotherapy as scheduled and improves safety and tolerability of HDMTX given with LV

ELIGIBILITY:
Inclusion Criteria:

* osteosarcoma
* eligible to receive 2 sequential cycles of HDMTX-LV

Exclusion Criteria:

* prior administration of glucarpidase
* progression of disease while on previous MTX treatment

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete Anderson, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Methotrexate Plus Glucarpidase Then Placebo: First cycle: High-dose methotrexate with leucovorin, plus 2 doses of glucarpidase 24 hours apart Second cycle: High-dose methotrexate with leucovorin, plus 2 doses of placebo 24 hours apart
- High-dose Methotrexate Plus Placebo Then Glucarpidase: First cycle: High-dose methotrexate with leucovorin, plus 2 doses of placebo 24 hours apart Second cycle: High-dose methotrexate with leucovorin, plus 2 doses of glucarpidase 24 hours apart
- Arm C, Compassionate Use of Glucarpidase: Compassionate use group to treat or prevent life threatening toxicity in the event of delayed elimination of MTX and/or renal impairment. Patients received glucarpidase 50 U/kg
Period: Overall Study
Arm/Group | High-dose Methotrexate Plus Glucarpidase Then Placebo | High-dose Methotrexate Plus Placebo Then Glucarpidase | Arm C, Compassionate Use of Glucarpidase
Started | 1 | 1 | 5
Completed | 1 | 1 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Methotrexate Plus Glucarpidase Then Placebo | High-dose Methotrexate Plus Placebo Then Glucarpidase | Arm C, Compassionate Use of Glucarpidase | Total
Number analyzed (Participants) | 1 | 1 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 3 | 5
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patients Progressing to Next Chemotherapy Cycle
Time Frame: 1 week after intervention
Arm/Group | High-dose Methotrexate Plus Glucarpidase Then Placebo | High-dose Methotrexate Plus Placebo Then Glucarpidase | Arm C, Compassionate Use of Glucarpidase
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | High-dose Methotrexate Plus Glucarpidase Then Placebo | High-dose Methotrexate Plus Placebo Then Glucarpidase | Arm C, Compassionate Use of Glucarpidase
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Methotrexate Plus Glucarpidase Then Placebo (N=1) | High-dose Methotrexate Plus Placebo Then Glucarpidase (N=1) | Arm C, Compassionate Use of Glucarpidase (N=5)
Febrile neutropenia (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 0 (0) | 1 (4)

LIMITATIONS AND CAVEATS:
No efficacy endpoints were reported due to early termination (insufficient enrollment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less